CLINICAL TRIAL: NCT02399748
Title: A Long-term Study for the Outcome of Pompe Disease
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200703045R
Record Dates: First submitted 2015-03-21; First posted 2015-03-26 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospectively follow patients with Pompe disease underwent enzyme replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

Confirm diagnosis with Pompe disease, is or is preparing receiving enzyme replacement therapy

Exclusion Criteria:

No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of Pompe disease who under enzyme replacement therapy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-04; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
all cause morbidities | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hsiu Chien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsu YK, Chien YH, Shinn-Forng Peng S, Hwu WL, Lee WT, Lee NC, Po-Yu Huang E, Weng WC. Evaluating brain white matter hyperintensity, IQ scores, and plasma neurofilament light chain concentration in early-treated patients with infantile-onset Pompe disease. Genet Med. 2023 Jan;25(1):27-36. doi: 10.1016/j.gim.2022.10.005. Epub 2022 Nov 18. PMID 36399131